CLINICAL TRIAL: NCT03129204
Title: Prevention of Post Intensive Care Syndrome in Family With SAF-T Intervention: Feasibility Study
Brief Title: Sensation Awareness Focused Training for Spouses
Acronym: SAF-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Paula Cairns, PhD, Principal Investigator, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00026246
Record Dates: First submitted 2017-02-08; First posted 2017-04-26 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Post Intensive Care Syndrome; Anxiety; Depression; Posttraumatic Stress Disorder; Sleep Deprivation
Keywords: intensive care unit; critical care; family; caregiver; actigraphy
MeSH Terms: conditions — postintensive care syndrome; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: prospective, randomized, experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAF-T Intervention Group (Experimental): The SĀF-T intervention includes coaching from SĀF-T trained research staff on awareness of biological sensations associated with events in the ICU that are perceived stressful. The research staff member will sit across from the participant and ask them to use their eyes to follow hand movements that will induce lateral left-right (saccadic) eye movements to elicit an orienting response that activates an investigatory reflex in which first, an alert response occurs and then, a reflexive pause produces decreased arousal in the face of no threat, which elicits a calming response that rapidly eliminates negative biological sensations of stress.
  Interventions: Behavioral: SAF-T
- Control Group (No Intervention): The control group will not receive the SAF-T intervention.

INTERVENTIONS:
Behavioral: SAF-T — The Rosenzweig Center for Rapid Recovery has recently developed an adaptation of their Accelerated Resolution Therapy (ART) for psychological trauma and depression, called Sensation Awareness Focused Training (SĀF-T), as an approach to rapidly eliminate negative biological sensations of stress. SĀF-T is designed to elicit a calming response; interrupt negative thoughts, negative feelings, and negative behaviors; and ultimately serve as a self-management stress reduction tool for individuals.
  Arms: SAF-T Intervention Group

SUMMARY:
The purpose of the feasibility study is prevention of Post Intensive Care Syndrome in Family (PICS-F), specifically in spouses of critically ill, mechanically ventilated patients, using a nonpharmacological intervention called Sensation Awareness Focused Training (SĀF-T). This will be accomplished using a prospective, randomized, experimental design to achieve robust and unbiased results.

DETAILED DESCRIPTION:
More than 5.7 million patients are admitted to intensive care units (ICU) each year in the United States. The technologically advanced ICU is an unfamiliar frightening environment to patients and their families. Critical illness is a family crisis. There is strong evidence that family distress in response to critical illness does not disappear after ICU discharge. The Society of Critical Care Medicine has identified a cluster of complications that occur in family members of ICU patients as Post Intensive Care Syndrome-Family (PICS-F). PICS in family members of adult ICU survivors includes symptoms of ongoing anxiety, depression, and post-traumatic stress disorder (PTSD). Data suggest that 70% of family members have symptoms of anxiety and 33% have symptoms of depression and PTSD, which can persist for ≥4 years. Moreover, symptoms of anxiety, depression, and PTSD are higher and persist longer in family members than in adult ICU survivors. Because PICS-F occurs with greater frequency in spouses and surrogate health decision-makers, this study will focus on participants whom are spouses of mechanically ventilated critically ill adults (typically sedated and unable to make health decisions).

To date, the focus of PICS-F research has been on description, detection, and prevalence of PICS-F. The approach in the proposed project focuses on prevention of PICS-F using an innovative rapid stress reduction intervention. The Rosenzweig Center for Rapid Recovery has recently developed an adaptation of their Accelerated Resolution Therapy (ART) for psychological trauma and depression, called Sensation Awareness Focused Training (SĀF-T), as an approach to rapidly eliminate negative biological sensations of stress. SĀF-T is designed to elicit a calming response; interrupt negative thoughts, negative feelings, and negative behaviors; and ultimately serve as a self-management stress reduction method for individuals. Lateral left-right (saccadic) eye movements are used to elicit an orienting response that activates an investigatory reflex in which first, an alert response occurs and then, a reflexive pause produces decreased arousal in the face of no threat, which elicits a calming response that rapidly eliminates negative biological sensations of stress. This response process is consistent with behavior of interpretation or reaction to challenge in McEwen's Allostasis Stress Theory. The investigators expect the SĀF-T intervention will enable spouses to better manage stress and reduce risk of PICS-F.

Sleep deprivation has been self-reported as one of the top stressors of family members of ICU patients. Sleep adequacy is defined as a combination of three factors: latency (the time it takes to fall asleep), efficiency ([time spent sleeping ÷ total time in bed] × 100), and duration of sleep. According to the American Academy of Sleep Medicine for adequate sleep, persons should fall asleep within 15 minutes, stay asleep for at least 85% of the time they are in bed, and have a total sleep time of no less than 7 hours. Reasons reported by family members for sleep deprivation include anxiety, tension, and fear. Sleep deprivation may play a role in the development of PICS-F. Although anxiety, tension, and fear are to be expected when a family member is critically ill, acknowledging these feelings and practicing relaxation techniques can reduce the impact that the feelings have on sleep. Therefore, management of stress in spouses throughout the daytime may also improve nighttime sleep/rest and further reduce risk of PICS-F.

ELIGIBILITY:
Inclusion Criteria:

* spouse of a critically ill, mechanically ventilated patient
* within 36 hours of admission to adult Tampa General Hospital (TGH) ICUs
* understands English

Exclusion Criteria:

* anticipation by the clinical provider of imminent patient death
* spouse does not understand English
* spouse is under the age of 18 years old
* spouse is currently receiving treatment for an existing PICS condition (anxiety, depression or PTSD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-03 (Actual); Primary Completion 2018-02-26 (Actual); Study Completion 2018-02-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Symptoms of Anxiety following ICU discharge and at 1 and 3 months post hospital discharge | Four time points: 1) upon study enrollment, 2) at least 24 hours post ICU discharge, 3) 1 month post hospital discharge, and 4) 3 months post hospital discharge.
  Hospital Anxiety and Depression Scale
Change from Baseline Symptoms of Depression following ICU discharge and at 1 and 3 months post hospital discharge | Four time points: 1) upon study enrollment, 2) at least 24 hours post ICU discharge, 3) 1 month post hospital discharge, and 4) 3 months post hospital discharge.
  Hospital Anxiety and Depression Scale
Change from Baseline Symptoms of Post Traumatic Stress Disorder following ICU discharge and at 1 and 3 months post hospital discharge | Four time points: 1) upon study enrollment, 2) at least 24 hours post ICU discharge, 3) 1 month post hospital discharge, and 4) 3 months post hospital discharge.
  Impact Event Scale

SECONDARY OUTCOMES:
Sleep | Up to 3 days in the intensive care unit (ICU)
  Actiwatch wrist actigraphy
Change from Baseline Symptoms of Stress following ICU discharge and at 1 and 3 months post hospital discharge | Four time points: 1) upon study enrollment, 2) at least 24 hours post ICU discharge, 3) 1 month post hospital discharge, and 4) 3 months post hospital discharge.
  Perceived Stress Scale

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L Munro, PhD, Study Chair — University of South Florida
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT03129204/Prot_SAP_000.pdf